CLINICAL TRIAL: NCT01893996
Title: Adalimumab to Mitigate Cardiovascular Risk in RA Patients With Well-Controlled Joint Disease
Brief Title: Study of Adalimumab to Lower Cardiovascular Risk in RA Patients With Well Controlled Joint Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jonathan Graf (Other)
Collaborators: American College of Rheumatology Research and Education Foundation (Other); AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Graf, Associate Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-09816
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Disease
Keywords: rheumatoid; arthritis; cardiovascular; adalimumab; tnf; biologic
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases; Arthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab (Experimental): Active Study Drug is Adalimumab (Humira) which is FDA approved to treat rheumatoid arthritis since 2003.
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Placebo is inert and matches study drug, including the pre-filled syringe, and is supplied by Abbvie, the study drug manufacturer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — Patients will be randomized 1:1 to receive either adalimumab or placebo for the first 26 weeks of the trial, and then after a 26 week washout period, will be crossed over into the other arm (either placebo or adalimumab) for weeks 52-78.
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis patients are at increased risk of cardiovascular disease because of systemic inflammation that can persist even in patients with well-controlled joint disease. We hypothesize that adding an anti-tumor necrosis factor medication, adalimumab, to standard non-biologic therapy for rheumatoid arthritis will improve endothelial function (reduce cardiovascular risk) in these patients. The design of the trial is as follows: 18 month prospective, randomized, double-blind crossover trial comparing the addition of adalimumab to the addition of placebo. The primary endpoint is a change in endothelial cell function, as detected by brachial artery FMD, at 6 months of adalimumab treatment compared to 6 months of placebo.

DETAILED DESCRIPTION:
Excess mortality associated with RA is due largely to CVD that is not explained by traditional risk factors. Although articular manifestations usually dominate the clinical picture, RA is a systemic inflammatory disease, and systemic inflammation is the thought to be the underlying mechanism responsible for the increased CVD risk associated with RA. Because chronic inflammation can persist in treated RA patients with little or no clinically detectable joint inflammation, treatment to targets based largely on clinically measured joint activity may not adequately suppress the systemic inflammation associated with progression of atherosclerosis. The ACR recommends treatment to a therapeutic target of low disease activity as determined by standardized clinical assessments. We hypothesize that treated RA patients who have reached this ACR target of low disease activity nonetheless have persisting systemic inflammation that contributes to atherogenesis. We further hypothesize that acceleration of RA-directed therapy with systemic anti-inflammatory treatments (TNF inhibition) in patients with low disease activity will improve endothelial function, reduce vascular inflammation and improve the functionality of HDL particles, key biological features in the progression of atherosclerosis and its clinical manifestations.

Trial design: Prospective, randomized, double-blind crossover trial comparing the addition of adalimumab to the addition of placebo.

Study population: 60 RA patients on non-biological DMARDs with low disease activity as determined by a standardized clinical assessment (Disease Activity Score 28 joints [DAS28] < 3.2).

Primary endpoint: Primary endpoint is change in endothelial cell function, as detected by brachial artery FMD, at 6 months of adalimumab treatment compared to 6 months of placebo. We postulate that anti-TNF therapy with adalimumab will lead to an absolute increase of 2% in FMD, which typically translates into a 15% reduction in cardiovascular event rates.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able and willing to give written informed consent and comply with the requirements of the study protocol.
* Diagnosis of Rheumatoid Arthritis by ACR 1987 or ACR/EULAR 2010 criteria.
* Low RA disease activity as defined by DAS28 < 3.2
* No anti-TNF medication or other biologic agent (abatacept, rituximab, or tocilizumab) within the 12 months prior to enrollment.
* If taking methotrexate, then on a stable dose between 7.5 mg and 25 mg (PO or SQ) weekly for at least 3 months prior to randomization. If on a DMARD other than methotrexate, then that DMARD must be at a stable therapeutic dose for at least 3 months prior to randomization.
* If taking prednisone, then a stable dose of less than or equal to 10 mg/daily for at least 1 month prior to randomization
* If NSAID taken on a regular, daily schedule, then patient must be on a stable dose for one week prior to FMD studies. PRN use is excluded within 1 week of FMD studies.
* Age > 18
* Subject must be able and willing to self-administer SQ injections or have available qualified person(s) or caregiver to administer SQ injections
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment
* Adequate renal function as indicated by serum creatinine < 2.0.
* No use of phosphodiesterase type 5 inhibitors (PDE5) (i.e. sildenafil, tadalafil, and vardenafil) 1 week prior to the study and during the course of the study.

Exclusion Criteria:

* Use of an anti-TNF or other biologic medication (Including but not limited to abatacept, rituximab, or tocilizumab) within the previous 12 months.
* Prior history of MI, CVA, CABG, PTCA, or peripheral vascular disease
* SBP > 140/90 at two months prior to study enrollment
* Diabetes mellitus requiring insulin therapy
* The following laboratory parameters at the Screening visit

  * Neutropenia (absolute neutrophil count < 1,500/microliter [ L]);
  * Thrombocytopenia (platelets < 100,000/ L);
  * Anemia (hemoglobin < 8 g/dL);
  * Greater than or equal to 3 times the upper limit of normal (ULN) for either of the following liver function tests (LFTs): aspartate transaminase (AST) or alanine transaminase (ALT);
  * Renal insufficiency (serum creatinine> 2.0 mg/dL)
* Purified protein derivative (PPD) test of > 5 mm induration regardless of prior BacilleCalmette Guerin vaccine administration or positive QuantiFERON®-TB Gold In-Tube Test (QFT-G_IT) without documentation of completed treatment or evidence of ongoing treatment of latent tuberculosis (TB) for 30 days. Subjects with active TB infection are excluded.
* History of positive PPD, positive QuantiFERON®-TB Gold In-Tube Test (QFT-G_IT), or chest x-ray findings indicative of prior TB infection, without documentation of either treatment for TB infection or chemoprophylaxis for TB exposure
* Prednisone dose > 10 mg/day (or equivalent dose of another corticosteroid) within 1 month of randomization
* Presence of open leg ulcers
* Chronic or persistent infection including but not limited to human immunodeficiency virus [HIV],hepatitis B, hepatitis C, listeriosis, TB, or other opportunistic infection)
* Active infection or severe infections requiring hospitalization or treatment with intravenous(IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to randomization, or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to randomization
* Receipt of a live vaccine within 4 weeks prior to randomization
* History of malignancy within the past 5 years other than treated localized carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma
* Any medical condition, such as uncontrolled diabetes with documented history of recurrent infections, unstable ischemic heart disease, known coronary artery disease or known significant cardiac arrhythmias or severe congestive heart failure (New York Heart Association classes III or IV), recent cerebrovascular accidents, severe, progressive or uncontrolled neurological disease, and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol
* Women of childbearing potential who are sexually active and who do not agree to practiceone of the following methods of contraception during the duration of the study

  * condoms, sponge, foams, jellies, diaphragm or intrauterine device;
  * oral or parenteral contraceptives for 2 months prior to study product administration;
  * a vasectomized partner;
  * abstinence
* Pregnant (all women of childbearing potential must have a negative serum pregnancy test) or breastfeeding
* Any investigational agent within the earlier of 4 weeks or 5 half-lives prior to randomization
* History of drug or alcohol abuse within 6 months prior to randomization
* Known allergy or hypersensitivity to any study products
* Any psychiatric disorder that prevents the subject from providing informed consent
* Inability or unwillingness to follow the protocol
* Any condition or treatment, which in the opinion of the investigator, places the subject at an unacceptable risk as a participant in the trial
* Any individual who plans to start or stop or change the dose of lipid lowering medication,antihypertensive medication, NSAIDS, Cox-2 inhibitors, aspirin within 1 month of the study or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Function | Weeks 0, 13, 26, 52, 65, 78
  The primary endpoint is the change in endothelial cell function, as detected by brachial artery flow-mediated dilitation.

SECONDARY OUTCOMES:
Change in vascular inflammation | Weeks 0 and 26
  Vascular inflammation at select body sites will be quantified by 18F-fluorodeoxyglucose positron emission tomography (FDG-PET).

OTHER OUTCOMES:
Improvement in HDL function | Weeks 0,26,52,78
  HDL function will be assessed by the ability of HDL to promote cholesterol efflux, to prevent low-density lipoprotein (LDL) oxidation and to express higher activity of paraoxonase, an antioxidant enzyme.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Graf, MD, Principal Investigator — University of California, San Francisco; Peter Ganz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco/San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- See also: UCSF Division of Rheumatology: Clinical & Epidemiological Research — https://rheumatology.ucsf.edu/research/clinical-epidemiological-research